CLINICAL TRIAL: NCT02890095
Title: Prospective, Multicenter, Epidemiological Case-control Study, to Establish a Possible Correlation Between Persistent Chemical Contaminants (POPs) and Breast Cancer.
Brief Title: Persistent Organic Pollutants and Breast Cancers (POPCASE)
Acronym: POPCASE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-N-2014-08
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A = Breast Cancer surgery (Experimental): Arm A : women undergoing breast cancer surgery.
  Interventions: Procedure: Breast cancer surgery
- Arm B = Control (plastic surgery) (Other): Arm B : women undergoing breast surgery for the purpose of plastic surgery
  Interventions: Procedure: plastic surgery

INTERVENTIONS:
Procedure: Breast cancer surgery — First, 2 specific adipose tissue samples will be performed during the surgery :
  * 1 sample near the tumor, to measure the contaminants (dioxins, PCBs, organochlorine pesticides, polybrominated compounds)
  * 1 remote sample of the tumor bed, superficial, at least 5 cm from the tumor, to be used to determine the level of expression of hormone receptors and to establish the expression profiles, after cutting and inclusion in paraffin blocks for marking IHC.
  These withdrawals are made during surgery, during surgery, as part of the intervention and the remodeling of the mammary gland (standard care for patients). This is unused balance for diagnostic.
  Before anaesthesia : specific blood samples (for the determination of circulating pollutants and for the analysis of gene polymorphism)
  Arms: Arm A = Breast Cancer surgery
Procedure: plastic surgery — The excision piece will follow the classical pathological circuit.
  A specific charge of subcutaneous adipose tissue will be performed as part of research on the surgical specimen. This sample will be used:
  * measuring contaminants (dioxins, PCBs, organochlorine pesticides, polybrominated compounds)
  * to determine the level of expression of hormone receptors and to establish the expression profiles, after cutting and inclusion in paraffin blocks for marking IHC. These samples are all made during surgery, for usual care surgery these patients.
  Before anaesthesia : specific blood samples (for the determination of circulating pollutants and for the analysis of gene polymorphism)
  Arms: Arm B = Control (plastic surgery)

SUMMARY:
Exposure to certain classes of chemical contaminants, including certain persistent organic pollutants (POPs) with a character of endocrine disruptors, could be one of the factors that lead to increase incidence of breast cancer in the Western world .

However, the causal role of POPs in the onset of breast cancer remains nowadays unproven. Preliminary epidemiological studies on the impact of these environmental factors in breast cancer etiology have ignored the critical periods of exposure. Similarly, they have considered a limited number of pollutants (not including possible joint or synergistic effects between individual compounds) and did not distinguish the different breast cancer subtypes may have different etiologies or even of genetic susceptibility factors (POP polymorphism of detoxification enzymes).

Thus, POPCASE study examines the association between the presence of breast cancer and the levels and exposure profiles to a group of POPs measured in adipose tissue (AT) and blood, in particular using spectrometric methods developed by the team LABERCA (Nantes, France). These internal levels of POPs (organochlorine pesticides, dioxins, PCBs, brominated flame retardants) will be measured both quantitatively (tissue concentrations) and qualitative (relative proportions of different pollutants sought).

DETAILED DESCRIPTION:
Exposure to certain classes of chemical contaminants, including certain persistent organic pollutants (POPs) with a character of endocrine disruptors, could be one of the factors that lead to increase incidence of breast cancer in the Western world .

However, the causal role of POPs in the onset of breast cancer remains nowadays unproven. Preliminary epidemiological studies on the impact of these environmental factors in breast cancer etiology have ignored the critical periods of exposure. Similarly, they have considered a limited number of pollutants (not including possible joint or synergistic effects between individual compounds) and did not distinguish the different breast cancer subtypes may have different etiologies or even of genetic susceptibility factors (POP polymorphism of detoxification enzymes).

Finally, this demonstration has not been done for 2 reasons:

* Multidisciplinary Issues,
* Need innovative tools for statistical analysis and interpretation of these more integrated environmental data.

Thus, POPCASE study examines the association between the presence of breast cancer and the levels and exposure profiles to a group of POPs measured in adipose tissue (AT) and blood, in particular using spectrometric methods developed by the team LABERCA (Nantes, France). These internal levels of POPs (organochlorine pesticides, dioxins, PCBs, brominated flame retardants) will be measured both quantitatively (tissue concentrations) and qualitative (relative proportions of different pollutants sought).

It is therefore to improve the level of knowledge between environmental chemical exposure and increased incidence of breast cancer (in its environmental, genetic and molecular components) within the general population, in response to a public health issue, the question of the actual impact on the health of major classes of chemical pollutants present in our environment and our staying power behind debates and being associated with high stakes, both scientists but economic and societal.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 and <75 years
2. According to the arm:

   * Arm A: histologically confirmed diagnosis of invasive breast cancer (only), unilateral or bilateral, outside off recurrence and relapse. Patients who have been supported for a contralateral breast cancer can be included if a period of at least 2-years between the last systemic treatment of inclusion in the study.
   * Arm B: Any woman operated on for breast plastic surgery (breast lift and breast reduction cure only)
3. Performance status (WHO) ≤ 1

5. Patient affiliated to a social security scheme, 6. Patient who signed and dated informed consent form 7. Arm A only: unifocal lesion 8. Arm A only: Clinical stage M0

Exclusion Criteria:

1. Patient with uncontrolled infection
2. Patient pregnant or lactating
3. Patient with a viral infection (HIV, Hepatitis B, Hepatitis C)
4. Patient cannot be regularly monitored for psychological reasons, social, family or geographical.
5. Patient Private of liberty or under a guardianship authority / curatorship.
6. Arm A only: Patient to benefit from neoadjuvant therapy for breast cancer
7. Arm A only Patient with metastatic breast cancer
8. Arm A only Patient diagnosed cancer in situ (intra ductal)
9. Arm A only Patient with BRCA1 or BRCA2 known
10. Arm B only: previous breast plastic surgery, regardless of the type of intervention

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
correlation between the individual risk of breast cancer and persistent chemical contaminants | 10 years after surgery
  The main objective is to establish a correlation between the individual risk of breast cancer and persistent chemical contaminants (POPs) respectively measured in adipose tissue (i.e. storage compartment) and blood (i.e. circulating compartment).
  => Comparison of the assay in the body of a set of chemical pollutants in the environment between the following two groups:
  * Group A: women receiving breast cancer surgery,
  * Group B: women receiving breast surgery for the purpose of plastic surgery (control) This contamination profile is "exposure of interest" in this study. The quantification of this exposure is based on a targeted measure, by mass spectrometry, an expanded set of representative substances of the main families of lipophilic POPs (pesticides, PCBs, dioxins and polybrominated compounds) present to trace (femtomol).

CONTACTS AND LOCATIONS:
Overall Officials: Mario CAMPONE, MD, PhD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (3):
- France (3):
  - Clinique Breteche, Nantes
  - ICO René Gauducheau, Saint-Herblain
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No